CLINICAL TRIAL: NCT03843606
Title: Modified Ketogenic Diet in Patients With McArdle Disease Part A - a Pilot Study
Brief Title: Modified Ketogenic Diet in Patients With McArdle Disease Part A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nicoline Løkken, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18013022
Record Dates: First submitted 2018-12-12; First posted 2019-02-18 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: McArdle Disease
MeSH Terms: conditions — Glycogen Storage Disease Type V

STUDY DESIGN:
Intervention Model Description: Open interventional study to investigate the effects of 3 different ketogenic diet regimes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diet 1 (Experimental): 60% fat, 15% protein, 25% carbohydrates
  Interventions: Other: Modified ketogenic diets
- diet 2 (Experimental): 70% fat, 15% protein, 15% carbohydrates
  Interventions: Other: Modified ketogenic diets
- diet 3 (Experimental): 80% fat, 15% protein, 5% carbohydrates
  Interventions: Other: Modified ketogenic diets

INTERVENTIONS:
Other: Modified ketogenic diets — Different diet composition

SUMMARY:
McArdle disease, glycogen storage disease type V, is a rare metabolic disease. Affected individuals are unable to utilize sugar stored as glycogen in muscle.

We hypothesize that a modified ketogenic diet could be a potential treatment option, by providing ketones as alternative fuel substrates for working muscle.

In this open interventional pilot study we wish to investigate 3 different modified ketogenic diet regimes, to find an optimal composition of a modified ketogenic diet that ensures adequate degree of ketosis and at the same time is well tolerated for patients with McArdle disease.

DETAILED DESCRIPTION:
Open interventional study to investigate 3 different modified ketogenic diet regimes, to find an optimal composition of a modified ketogenic diet for patients with McArdle disease

McArdle disease, glycogen storage disease type V, is a rare metabolic disease caused by mutations in the PYGM gene resulting in absence of the enzyme muscle phosphorylase. Affected individuals are unable to utilize sugar stored as glycogen in muscle, leading to exercise intolerance, exercise-induced muscle pain, contractures and rhabdomyolysis, which may cause renal failure. Currently, there are no satisfactory treatment options for McArdle disease. Ketones are feasible fuel alternatives to muscle glycogen when muscle glycogenolysis is blocked as in McArdle disease.

A key element of alleviating symptoms in McArdle disease is to provide alternative fuels for energy metabolism. Ketosis can potentially provide alternative fuel substrates by provision of endogenous ketone bodies (KBs) which are desirable fuels for skeletal muscle and brain. Ketosis can be reached by fasting and can be induced by adhering to a modified ketogenic diet, which entails a high-fat, low-carbohydrate diet, which simulates the metabolic effects of fasting.

The optimal modified ketogenic diet composition, that ensures adequate degree of ketosis and at the same time is well tolerated, has not been investigated in patients with McArdle disease. Therefore this pilot study seeks to investigate which of 3 different diets is the most optimal ad effective for patients with McArdle disease. The 3 different diets will have carbohydrate percentages ranging from 5-25%, and fat percentage from 60-80%.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed GSDV
* Patient is willing and able to provide written informed consent prior to participation.
* Patient is ambulatory.
* Women in fertile age must be willing to practice the following medically acceptable methods of birth control

Exclusion Criteria:

* Patient has any prior or current medical conditions that, in the judgment of the Investigator, would prevent the patient from safely participating in and/or completing all study requirements.
* Pregnancy or breastfeeding
* Patient does not have the cognitive capacity to understand/comprehend and complete all study assessments
* Patients with porphyria or disorders of fat metabolism (primary carnitine deficiency, carnitine palmitoyltransferase I or II, β-oxidation defects etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Heart rate | 2 times
  heart rate during constant load cycling exercise

SECONDARY OUTCOMES:
Compliance | 3 weeks
  Dietary diary to evaluate compliance and diet acceptability
indirect calorimetry | 2 times
  Oxidation rates measured via indirect calorimetry during constant load cycling calorimetry
level of ketosis | daily
  Ketone bodies in the blood
Safety parameters | 2 times
  Blood samples
Perceived exertion | 2 times
  Borg scale during constant load cycling
other blood samples | 2 times
  Cholesterol, fatty acids, hormones, ammonia

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No